CLINICAL TRIAL: NCT04690257
Title: The Effectiveness of Art Therapy on Reducing Pain and Anxiety in Children Receiving Venipuncture in a Pediatric Department: A Randomized Controlled Trial
Brief Title: Effectiveness of Art Therapy on Reducing Pain and Anxiety in Children Receiving Venipuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Sherzad Khudeida Suleman, Principal Investigator (PhD Student), University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SSKhudeida
Record Dates: First submitted 2020-12-26; First posted 2020-12-30 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Venipuncture; Pain; Anxiety; Fear
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TICK-B group as Intervention group (Experimental): Experimental: TICK-B group
  -Pediatric patients received TICK-B as a distraction in the TICK-B group
  Interventions: Other: Trace Image and Coloring for Kids-Book (TICK-B)
- Standard care provided group as control group (No Intervention): -Pediatric patients received standard care (routine care) in the control group.

INTERVENTIONS:
Other: Trace Image and Coloring for Kids-Book (TICK-B) — A collection of pictures designed as a book contains and given to children during the procedure and they take a picture as they favored.
  Arms: TICK-B group as Intervention group

SUMMARY:
Venipuncture is one of the most common stressful procedures in children. Managing pain and fear of venipuncture procedure recommended strongly because it may change children's memory for procedural pain and the subsequent acceptance of later health care painful interventions. Prior painful experiences can reduce the acceptance of later health care, hence making it more difficult for both patients and nurses.

There was clear evidence that the distraction method is the most performed as a psychological technique performed to decrease venipuncture-related pain and distress and supporting its efficacy in children.

The aim of this study to investigate the effectiveness of TICK-B on children's pain and anxiety during venipuncture procedure.

DETAILED DESCRIPTION:
Note:

The first registration number for the protocol of Ph.D. was approved as 10092019-6 on 10th September 2019 It approved the grant to publish the result as 20072020-3 on 23, August,

ELIGIBILITY:
Inclusion Criteria:

* being between 6-12 years old,
* a physician order was placed for the blood sample,

Exclusion Criteria:

* Chronic medical condition.
* Those whose parent not participated,
* Neurodevelopmental delayed, verbal difficulties, difficulties in hearing or visual,
* Unconsciousness.
* Take a medication analgesic in the past 6 hrs.
* history of syncope.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Measure | Immediately after venipuncture (1-2 min)
  Wong-Baker faces scale (WBFS). Used to measure the pain severity during the procedure, the WB-FBRS is a series of six cartoon faces positioned side-by-side from the greatest pain to the mildest one (0-5).

SECONDARY OUTCOMES:
Fear Measure | Immediately after venipuncture (1-2 min. )
  The Childrens Fear Scale (CFS) is used to assess children's fear or anxiety levels. The one-item scale consists of five sex neutral faces arranged from left to right with no fear in the center, through fear out to extreme fear.

OTHER OUTCOMES:
Pain and anxiety measured by parents and observe. | Immediately after venipuncture (1-2 min.)
  Visual Analog Scale (VAS) was used to measure the pain and fear of children by parents and observer. A rating of 0 represents no pain and 10 represents the worst or most severe pain. The VAS is a valid, reliable, and frequently used measure of procedural distress in children 6 to 18 years of age.

CONTACTS AND LOCATIONS:
Overall Officials: Akram M Atrushi, Professor, Study Chair — Duhok University; Margareta Halek, Professor, Study Director — Witten\Herdecke University
Locations (1):
- Sherzad Suleman, Witten, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suleman SK, Atrushi A, Enskar K. Effectiveness of art-based distraction on reducing pediatric patients' pain and anxiety during venipuncture: A randomized controlled trial. Complement Ther Clin Pract. 2022 Aug;48:101597. doi: 10.1016/j.ctcp.2022.101597. Epub 2022 Apr 30. PMID 35512482